CLINICAL TRIAL: NCT04619771
Title: M-Health Administered Sleep Treatment to Enhance Recovery in Bariatric Populations (MASTER)
Acronym: MASTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Johns Hopkins University (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Genna Popovich Hymowitz, Clinical Assistant Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2020-00283
Record Dates: First submitted 2020-10-27; First posted 2020-11-06 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Insomnia; Morbid Obesity
Keywords: Insomnia; Sleep; Bariatric Surgery; Morbid Obesity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Obesity, Morbid | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy for Insomnia (Experimental): CBT-I has a specific protocol with behavioral targets that differ significantly from standard CBT. This approach focuses on implementing sleep restriction and stimulus control interventions which are fully deployed during the first session. We will deliver 5 CBT-I sessions over the course of 8 weeks. Key recommendations include: 1) reduce time in bed; 2) get up at the same time every day; 3) do not go to bed unless sleepy; 4) do not stay in bed awake for more than 15 minutes; and 5) avoid napping. Participants are also taught relaxation strategies and cognitive therapy addresses arousal and catastrophizing.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — CBT-I has a specific protocol with behavioral targets that differ significantly from standard CBT. This approach focuses on implementing sleep restriction and stimulus control interventions which are fully deployed during the first session. 5 CBT-I sessions will be delivered over the course of 8 weeks. Key recommendations include: 1) reduce time in bed; 2) get up at the same time every day; 3) do not go to bed unless sleepy; 4) do not stay in bed awake for more than 15 minutes; and 5) avoid napping. Participants are also taught relaxation strategies and cognitive therapy addresses arousal and catastrophizing.
  Other Names: CBT-I

SUMMARY:
This study is a longitudinal clinical trial designed to assess the feasibility of sleep intervention (Cognitive Behavioral Therapy for Insomnia (CBT-I)) in individuals with insomnia following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Fluency with English
* Willingness to maintain an active telehealth platform account
* Daily access to wireless internet connection or sufficient cell phone service for telemedicine
* Undergone bariatric surgery (Roux-en-Y or vertical sleeve gastrectomy) within past 1-3 years
* Must have experienced <50% excess weight loss following surgery Clinically significant insomnia (i.e., ISI score >11)

Exclusion Criteria:

* Patient underwent revision of initial weight loss procedure
* PHQ-9 Depression score > 15
* GAD-7 Anxiety score > 15
* Current alcohol or substance abuse
* Current narcotic use
* Unstable major psychiatric condition
* Restless leg syndrome
* Sleep apnea with non-adherence to CPAP intervention (i.e., use of CPAP <4 nights/week)
* Other problems at investigator discretion
* Vulnerable populations (e.g., adults unable to consent, ages <18, pregnant women, and prisoners).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Follow Up (week 15)
  Number of participants screened into the study per month will help measure feasibility.
Completion of Study Measures | Follow Up (week 15)
  The average percentage of study measures (self-report questionnaires, daily diaries and CBT-I sessions) that are completed across participants will help determine feasibility.
ActiGraph Use | Follow Up (week 15)
  The average percentage of days spent wearing the medical-grade Fitbit-like-device that collects sleep and physical activity data to help assess feasibility.
Actigraph Compliance | Follow Up (week 15)
  The average percentage of hours of wear per day of the medical-grade Fitbit-like-device that collects sleep and physical activity data to help assess feasibility.

SECONDARY OUTCOMES:
Treatment Acceptability | Follow Up (week 15)
  Treatment Acceptability Questionnaire will measure acceptability with patient-reported treatment satisfaction, and open-ended questions about satisfaction with both CBT-I and telemedicine (e.g., "What did you think about treating sleep as part of your Bariatric care?"; "How did you feel about getting treatment without being face-to-face?"; "What could we do to improve your treatment experience?").
Change in sleep onset latency | Follow-up (week 15)
  Sleep parameters will be measured by the ActiGraph model wGT3X-BT, a wrist-accelerometer.
Change in wake after sleep onset (WASO) | Follow-up (week 15)
  Sleep parameters will be measured by the ActiGraph model wGT3X-BT, a wrist-accelerometer.
Change in total sleep time (TST) | Follow-up (week 15)
  Sleep parameters will be measured by the ActiGraph model wGT3X-BT, a wrist-accelerometer.
Change in sleep efficiency | Follow-up (week 15)
  This will be measured by actigraph data and data from participant daily sleep logs.
Change in Insomnia Severity | Visit 1 (Week 3), Visit 5 (Week 11), Follow up (Week 15)
  The Insomnia Severity Index will be used to assess insomnia symptoms. The total score ranges from 0 to 63, with higher scores indicating more severe insomnia symptoms.
% Excess Weight Loss | Baseline (week 1), Follow-up (week 15)
  Measured weight data will be extracted from electronic medical records. The following formula will be used to calculate % excess weight loss. %EWL = [(Initial Weight) - (Post Intervention Weight)] / [(Initial Weight) - (Ideal Weight)]. Ideal weight will be extracted from the EMR.
Change in BMI | Baseline (week 1), Follow-up (week 15)
  BMI will be extracted from electronic medical records and the formula: ΔBMI = (Initial BMI) - (BMI at week 15) will be used to calculate change in BMI.
% Total Weight Loss | Baseline (week 1), Follow-up (week 15)
  Weight data will be extracted from the electronic medical record. %TWL will be calculated using the following formula: % TWL= [(Initial Weight) - (Post intervention Weight)] / [(Initial Weight)]× 100

CONTACTS AND LOCATIONS:
Overall Officials: Genna F Popovich Hymowitz, Ph.D., Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No